CLINICAL TRIAL: NCT05900310
Title: Retrospective Validation Study of Clinical Decision Support (CDS) Recommendations in the Linus Health Core Cognitive Evaluation
Brief Title: Linus Health CDS Retrospective Validation Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Linus Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CDSV-001
Record Dates: First submitted 2023-05-31; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Cognitive Impairment; Motor Disorders; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Motor Disorders; Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Core Cognitive Evaluation (CCE) — The Linus Health Core Cognitive Evaluation (CCE) is an easy-to-use but powerful tool to augment and facilitate cognitive health assessment during a patient's visit to their PCP. As a digital assessment solution, the CCE combines objective insights into cognitive ability with patient-reported insights to detect early signs of cognitive impairment and reveal specific modifiable risk factors earlier than the existing status quo assessments. The CCE is an FDA-listed Class II 510k exempt software as a medical device. The CCE has two components: The Digital Clock and Recall (DCR™) test and the Life and Health Questionnaire (LHQ).

SUMMARY:
This study is a retrospective validation study of deidentified Clinical Decision Support (CDS) recommendations generated by the Linus Health Core Cognitive Evaluation (CCE) for patients who have completed the CCE.

Site investigators consist of clinical experts including neurologists and geriatricians in the U.S. After signing the study agreements, the experts will receive batches of anonymized CCE outputs of patients and will rate the appropriateness of each CDS recommendation for each patient based on their review of the CCE results and their clinical judgment and expertise. The experts will also rate the clinical appropriateness of various parts of CDS pathways that form the LH CDS decision tree.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 and above
* Has already completed the Linus Health CCE

Exclusion Criteria:

* Incomplete CCEs
* CCEs that are flagged as "Requires clinician review"

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 55 and above, with or without cognitive symptoms, across all the healthcare organizations that Linus Health has been deployed in.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Median rating of each CDS recommendation | 2-3 weeks
  Rating of clinical appropriateness on the scale of 1 (extremely inappropriate) to 9 (extremely appropriate) for each set of CDS recommendations generated by the Linus Health CCE.

SECONDARY OUTCOMES:
Intraclass correlation coefficient (ICC) of each rating | 2-3 weeks
  ICC of each rating of clinical appropriateness to evaluate the inter-rater variability.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Jannati, MD, PhD, Principal Investigator — Linus Health
Locations (1):
- Linus Health, Inc., Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No